CLINICAL TRIAL: NCT00723216
Title: Multicenter, Randomized, Open-label Study to Evaluate the Efficacy and Safety of Enoxaparin Sodium (RP54563) 20mg Bid for 14 Days for Prevention of Venous Thromboembolism in Patients With Curative Abdominal Cancer Surgery. Physical Prophylaxis Only Arm [Intermittent Pneumatic Compression (IPC)] Will be Used as an Indicator of Event Rates.
Brief Title: Japanese Efficacy and Safety Study of Enoxaparin in Patients With Curative Abdominal Cancer Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: International Clinical Development, Study Director, Sanofi-aventis
Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EFC10094
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2010-04-05 (Estimated); Status verified 2010-04

CONDITIONS: Abdominal Neoplasms
Keywords: Prevention; venous thromboembolism; curative surgery
MeSH Terms: conditions — Abdominal Neoplasms; Venous Thromboembolism | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Enoxaparin
  Interventions: Drug: enoxaparin
- 2 (Other): Intermittent Pneumatic Compression (IPC)
  Interventions: Other: Physical prophylaxis

INTERVENTIONS:
Drug: enoxaparin — 20 mg twice a day
  Arms: 1
Other: Physical prophylaxis
  Arms: 2

SUMMARY:
The primary objective of this study is to evaluate the effects of enoxaparin on venous thromboembolism incidence and bleeding rate (major and minor bleeding) in patients undergoing curative abdominal cancer surgery. The secondary objective is evaluate the incidence of adverse events of enoxaparin in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Malignant tumor patients undergoing laparotomy for which surgery is expected to take 45 minutes or more.

Exclusion Criteria:

* surgery under laparoscope and other endoscopic operations
* clinical signs of deep vein thrombosis
* use of non-steroidal anti-inflammatory drugs from surgery completion until initial administration
* severe hepatic disease or renal disease
* women of childbearing potential, pregnant or lactating.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Venous thromboembolism incidence | 28 days

SECONDARY OUTCOMES:
Incidence of deep vein thrombosis, pulmonary thromboembolism, and venous thromboembolism incidence except patients with thrombus only in muscle veins, and incidence of proximal vein thrombosis | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: International Clinical Development, Clinical Study Director, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Tokyo, Japan